CLINICAL TRIAL: NCT06117553
Title: Clinical Study on the Application of Thorough Flushing Strategy During Colonoscopy Examination
Brief Title: Thorough Flushing Strategy During Colonoscopy Examination
Status: Completed | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zhao Hang, Head of Department of Gastroenterology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: KY-103-01
Record Dates: First submitted 2023-10-26; First posted 2023-11-07 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Colonoscopy
Keywords: colonoscopy, quality, polyps
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- limited: patients adopted limited flushing strategy
- thorough: Thorough flushing strategy
  Interventions: Procedure: thorough flushing

INTERVENTIONS:
Procedure: thorough flushing — The thorough flushing strategy refers to the thorough flushing of all liquid and foam accumulation areas during the inspection. Make all liquid accumulation parts in the intestinal cavity free of aspiratable liquid retention
  Groups: thorough

SUMMARY:
The investigators plan to adopt a thorough flushing strategy when withdrawing the endoscope, and have zero tolerance for the liquid and foam in the intestinal lumen. Observe and compare the impact of this strategy with traditional limited degree suction methods on the results of colonoscopy. The research group and the control group respectively adopted a thorough flushing strategy and a limited flushing strategy, and compared the total time of colonoscopy examination, the time of withdrawal, the detection rate of polyps, the detection rate of small polyps, and the amount of flushing fluid between the two groups. Analyze the value of thorough flushing strategy for the efficiency and quality of colonoscopy examination.

DETAILED DESCRIPTION:
Most physicians do not adopt a strategy of complete suction of fluid from the intestinal lumen during colonoscopy. There are both concerns about the time required for colonoscopy and the possibility of inability to thorough cleannig up. Some endoscopists believe that the visual field for partial cleaning of fecal water is acceptable and does not affect observation. This study aims to make an observation and comparison based on the existing problems mentioned above. With the help of direct water injection system, the investigators plan to adopt a thorough flushing strategy when withdrawing the endoscope, and have zero tolerance for the liquid and foam in the intestinal lumen. Observe and compare the impact of this strategy with traditional limited degree suction methods on the results of colonoscopy. The research group and the control group respectively adopted a thorough flushing strategy and a limited flushing strategy, and compared the total time of colonoscopy examination, the time of withdrawal, the detection rate of polyps, the detection rate of small polyps, and the amount of flushing fluid between the two groups. Analyze the value of thorough flushing strategy for the efficiency and quality of colonoscopy examination.

ELIGIBILITY:
Inclusion Criteria:

* People without contraindications for colonoscopy

Exclusion Criteria:

* Patients diagnosed with colon polyps

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 160 patients were selected for colonoscopy examination and randomly assigned to the study group and control group. The two groups used a thorough flushing strategy and a limited flushing strategy to complete colonoscopy examination. The research group adopted a thorough flushing strategy, while the control group adopted a limited flushing strategy. The thorough flushing strategy refers to the thorough flushing of all liquid and foam accumulation areas during the inspection. Make all the liquid accumulation parts in the intestinal cavity free of aspiratable liquid retention. The limited flushing strategy refers to not pursuing full liquid suction, but flushing until it is clear enough for observation. The limited flushing strategy is currently the conventional flushing method for colonoscopy.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
time of examination | 1week
  the time from insertion to exit the anus
time of insertion | 1week
  the time from insertion to arriving at cecum
time of withdrawl | 1week
  the time from cecum to anus
number of polyps | 1week
  the number of polyps found
location of polyps | 1week
  the location of polyps found
shape of polyps | 1week
  the shape of polyps found, classified into lateral, senssile and pediculated three types

SECONDARY OUTCOMES:
Boston score | 1week
  the Boston score of bowel preparation (from 0-9)
volume of water | 1week
  volume of water used for flushing

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No